CLINICAL TRIAL: NCT05215782
Title: Evaluation of Optina Retina Scans to Detect the Likeley Cerebral Amyloid Status (CAS) as Determined by Prospective PET Imaging
Brief Title: Eye to Brain Connection
Status: Completed | Type: Observational
Sponsor: Optina Diagnostics Inc. (Industry)
Collaborators: Ezy Medical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: DOC100681
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-randomized, non-treatment, observational study designed to discover correlations between retinal imaging and amyloid PET imaging. Subjects will be recruited to the clinical cohort from referring physicians. Subjects may be participants from existing studies and clinical practices

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 50 to 90 years (inclusive).
2. Individuals with reported cognitive complaint (self or from an informant) under clinical investigation by a health professional for cognitive impairment where Alzheimer's disease (AD) is one of the differential diagnoses.
3. Demonstrated cognitive impairment as evidenced by at least one of the following:

   1. Mini Mental State Examination (MMSE) score < 26/30
   2. Montreal Cognitive Assessment (MoCA) score < 26/30
   3. Score > 1 Standard Deviation below population mean on a standardized neuropsychological test, based on normative data from age-, sex-, education-, and where possible, race-matched peers [Based on guidelines for detecting Mild Cognitive Impairment due to AD (Albert et al., 2011)]
4. Cognitive impairment on the above test/s is unable to be fully explained by systemic, neurological or psychiatric disorders other than Alzheimer's disease.
5. Capacity to give informed consent by patient or Legally Authorized Representative (LAR).
6. Ability to undergo PET and MRI scans.

Exclusion Criteria:

1. Any ophthalmologic condition that would prevent obtaining retinal imaging and/or could interfere with the analysis of the MHRC-C1 images by the CAS, including:

   * Pupil dilation contraindicated (due to a pathology, or presence of 3 quadrants with Van Herick frading of 0 or 1 without iridotomy)
   * Inadequate pupil dilatation (< 6mm diameter) preventing uniform illumination of the retina with the MHRC-C1
   * Diagnosis of glaucoma or signs of glaucoma (excavation ratio ≥0.7)
   * Signs of vascular occlusion or retinopathy (microaneurysm, exudate, hemorrhage or edema) within a diameter of 10 mm from the mid-point between the optic nerve head and the macula
   * Presence of drusen and/or age-related macular degeneration (AREDS 9-step scale

     * 4 - cumulative drusen area diameter ≥ 250 um, pigmentary changes and cumulative drusen area diameter ≥ 63 um or pigmentary changes and cumulative geographic atrophy area diameter ≥ 354 um)
   * Macular anomaly (e.g. macular hole, dystrophy, degeneration)
   * Nuclear sclerosis > 2 (LOCS II four-point grading system) or presence of central cortical or central posterior subcapsular cataract
   * Deficient visual fixation (inability to fixate for at least 2 s)
   * Refractive error outside the range of -15 D to +15 D
   * Corneal or media opacities (e.g. Weiss ring) affecting retinal imaging on a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula (i.e. the area of interest for the MHRC-C1 imaging)
   * Scar, atrophy, naevus, tumor, epiretinal membrane or retinal pucker with a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula
   * Papilledema
2. Inability of obtaining at least 3 images of satisfactory quality with the MHRC-C1 per the Optina Diagnostics quality index software.
3. Impossibility of obtaining a satisfactory quality amyloid-PET scan for interpretation by imaging specialists.
4. Individuals currently enrolled in cerebral amyloid modifying medication studies.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 adults between 50 and 90 years old, and undergoing evaluation for Alzheimer's Disease or other cognitive impairments will be recruited from the community. Patients will be asked if they would like to hear about a study related to better diagnostic tools for cognitive decline and dementias, which is seeking volunteers to undergo a non-invasive eye scan with a new type of camera. Informed consent will be obtained prior to enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
To identify features in the retinal hyperspectral images that strongly correlate with the cerebral Aβ plaque status (positive or negative) measured with amyloid PET imaging. | 1 year

SECONDARY OUTCOMES:
Evaluate the classification performance of the Optina software to detect the likely cerebral amyloid status. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ezy medical research, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No